CLINICAL TRIAL: NCT03506009
Title: Argatroban Plus R-tPA for Acute Posterior Circulation Infarction (AR-PCI): a Prospective, Random, Blinded Assessment of Outcome and Open Label Multi-center Study
Brief Title: Argatroban Plus r-tPA for Posterior Circulation Infarction（AR-PCI）
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: it is very difficult to recruit qualified patients
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: k(2017)29
Record Dates: First submitted 2018-04-15; First posted 2018-04-23 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Argatroban, Rt-PA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Argatroban combined with rt-PA (Experimental)
  Interventions: Drug: Argatroban combined with rt-PA
- rt-PA (Active Comparator)
  Interventions: Drug: rt-PA

INTERVENTIONS:
Drug: Argatroban combined with rt-PA — Argatroban as a 100-ug/kg bolus over 3 to 5 minutes was administered intravenously within 1 hour of the tPA bolus followed by a continuous Argatroban infusion of 1.0 ug/kg per minute for 48 hours adjusted to a target activated partial thromboplastin time of 1.75 X baseline (about 10%).
  Arms: Argatroban combined with rt-PA
Drug: rt-PA — Intravenous throbolysis with 0.9mg/kg rtPA.
  Arms: rt-PA

SUMMARY:
Acute ischemic stroke (AIS) is the most common type of stroke, which has high rate of morbidity, mortality and disability. A large number of studies have confirmed that the thrombolytic therapy can effectively open blood vessels and improve the functional prognosis of acute ischemic stroke. Therefore, all guidelines recommend giving thrombolysis treatment to acute ischemic stroke patients within 4.5 hours of onset. However, about 1/3 patients receiving thrombolysis will have good prognosis, while a large number of patients will still be disabled and even dead. How to improve the neurofunction prognosis of thrombolytic patients has been a hot topic in the world.

Recent studies have found that the combined application of argatroban and rt-PA in the treatment of acute anterior circulation infarction might improve the clinical prognosis and not significantly increase bleeding. Some studies have reported that the combined application of argatroban and rt-PA could improve the blood vessel opening rate, and prevent re-occlusion after opening.

Based on the discussion, the present study is designed to explore the efficacy and safety of argatroban plus rt-PA in the treatment of acute posterior circulation infarction.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Diagnosis of posterior circulation ischemic stroke;
3. Time from onset to treatment ≤6 hours;
4. NIHSS: 4-25;
5. Signed informed consent by patient self or legally authorized representatives.

Exclusion Criteria:

1. mRS≥2;
2. History of stroke within 3 months;
3. History of intracranial hemorrhage;
4. Suspected subarachnoid hemorrhage;
5. Intracranial tumour, vascular malformation or arterial aneurysm;
6. Major surgery within 1 month;
7. Systolic pressure ≥180 mmHg or diastolic pressure ≥110 mmHg;
8. Platelet count < 105/mm3;
9. Heparin therapy or oral anticoagulation therapy within 48 hours;
10. Abnormal APTT;
11. Thrombin or Xa factor inhibitor;
12. Severe disease with a life expectancy of less than 3 months;
13. Blood glucose < 50 mg/dL (2.7mmol/L);
14. Patients who have received any other investigational drug or device within 3 months;
15. Pregnancy;
16. Researchers consider patients inappropriate to participate in the registry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Proportion of mRS (0-1） | 90±7 days

SECONDARY OUTCOMES:
Early neurological deterioration | 48 hours
  4 or more increase in NIHSS
Proportion of mRS (0-2） | 90±7 days
the occurence of stroke | 90±7 days
symptomatic intracranial hemorrhage | 36 hours

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China